CLINICAL TRIAL: NCT05095818
Title: Impact of Nursing Involvement on Implementation of Human Immunodeficiency Virus (HIV) Prevention Services in an Academic Obstetric/Gynecologic (OB/GYN) Clinical Setting
Brief Title: Impact of Nursing Involvement on Implementation of HIV Prevention Services
Acronym: PrEP-RN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00209380
Record Dates: First submitted 2021-10-13; First posted 2021-10-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pre-Exposure Prophylaxis (PrEP)

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care with EMR Enhancements (No Intervention): Participants in this arm will receive Standard of Care with EMR Enhancements.
- Standard of Care with EMR Enhancements and PrEP-RN (Experimental): Participants in this arm will receive Standard of Care with EMR Enhancements and PrEP-RN.
  Interventions: Other: PrEP-RN

INTERVENTIONS:
Other: PrEP-RN — Patients randomized to the intervention arm will be counseled on HIV risk factors in general, their HIV risk factors in particular, and prevention methods, inclusive of PrEP (Emtricitabine 200 mg/Tenofovir disoproxil fumarate 300 mg).
  Arms: Standard of Care with EMR Enhancements and PrEP-RN

SUMMARY:
Women comprise 20% of new Human Immunodeficiency Virus (HIV) diagnoses in the United States (U.S.) with 86% attributed to heterosexual contact. HIV pre-exposure prophylaxis (PrEP) uptake among cisgender women (women who are assigned female at birth and identify as women) is low.

A randomized controlled trial (RCT) will assess the feasibility and effectiveness of a registered nurse (RN)-led PrEP project in Obstetrics and Gynecology (OB/GYN) clinics. The PrEP-RN will counsel patients about their risks for HIV acquisition via telemedicine. Under protocol guidance, the PrEP-RN will order laboratory tests and initiate PrEP for at-risk women. A total of 440 at-risk cisgender women will be randomized 1:1 to the standard of care with electronic medical record (EMR) enhancements (e-SOC) or e-SOC with the PrEP-RN.

DETAILED DESCRIPTION:
This project will be launched in three OB/GYN outpatient clinics of a single academic medical system in Baltimore, Maryland. Baltimore City is one of the 57 jurisdictions targeted in the federal government's Ending the HIV Epidemic (EHE) Initiative.

To test the investigators' hypothesis that an RN can effectively counsel about PrEP, initiate therapy, and follow patients with minimal practitioner involvement, the investigators plan to conduct a randomized controlled trial with two arms. The control arm will include an enhanced standard of care (e-SOC), which is standard of care plus electronic medical record (EMR) changes. These EMR changes will include best practice alerts (BPAs) that encourage nurses and practitioners to add HIV risk-related codes to patients' problem lists, as well as order sets and note templates to facilitate PrEP initiation. The intervention arm will include the PrEP-RN plus e-SOC.

Patients randomized to the intervention arm will first be contacted via an electronic patient portal integrated with the EMR. While most of the investigators' patients utilize this patient portal, if a patient does not have access, this step will be skipped. Follow-up telephone calls will then be made to counsel patients on HIV risk factors in general, the patient's HIV risk factors in particular, and prevention methods, inclusive of PrEP. PrEP, including same-day PrEP, will be offered. If a patient declines PrEP, no additional attempts will be made by the PrEP-RN to counsel the patient.

If a patient decides to initiate PrEP, the PrEP-RN will place and order the required laboratory tests. The PrEP-RN will utilize the PrEP order set in the EMR to order labs, prescribe medication electronically to the patient's pharmacy, provide patient education, and schedule follow-up appointments. All orders and prescriptions will be sent to the clinic's Medical Director for authorization.

A Manual of Procedures was created for the PrEP-RN to carry out each step of PrEP initiation and follow-up. The manual outlines how to respond to abnormal tests, provide prescription coverage assistance, and coordinate care with other specialties as needed to address test results. The PrEP-RN will be responsible for follow-up visits and will contact the patients one-two weeks after medication initiation. At this time, the PrEP-RN will review the importance of daily adherence to PrEP and assess for any side effects.

If successful, our PrEP intervention could be implemented in other settings and largely improve current strategies for increasing PrEP utilization among at-risk cisgender women.

ELIGIBILITY:
Inclusion Criteria:

* not living with HIV
* weight >35 kg
* receiving OB/GYN care in our preselected clinics
* GYN patients: positive sexually transmitted infection (STI) diagnosis within past 6 months, or if seeking STI testing and a have a history of an STI
* OB patients: at least one positive answer to the following risk screen: inject illicit drugs; sex with a partner who injects illicit drugs; any past STIs; sex with a partner who has sex with both men and women; sex for money, drugs, other payment; sex with a partner currently infected with HIV; sex with more than one partner

Exclusion Criteria:

* symptoms or clinical signs consistent with acute HIV infection
* unknown HIV infection status
* allergies to the active substances or any excipients of PrEP
* estimated creatinine clearance of <60 mL/minute
* active Hepatitis B infection
* participating in other clinical studies related to HIV and/or antiretroviral therapy

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Assigned female at birth
Enrollment: 440 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
Awareness of PrEP as assessed by percentage of at-risk women who receive HIV risk prevention counseling | During the study interval, up to 16 months
  Awareness of PrEP will be assessed by the percentage of at-risk women with EMR documentation of HIV risk prevention counseling.

SECONDARY OUTCOMES:
Percentage of women at risk for HIV who initiate PrEP | During the study interval, up to 16 months
  Measured by the number of PrEP laboratory tests and the number of PrEP prescriptions ordered.

CONTACTS AND LOCATIONS:
Overall Officials: Jenell Coleman, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States